CLINICAL TRIAL: NCT02502253
Title: BDPP Treatment for Mild Cognitive Impairment (MCI) and Prediabetes or Type 2 Diabetes Mellitus (T2DM)
Acronym: BDPP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00062802
Record Dates: First submitted 2015-07-08; First posted 2015-07-20 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-06

CONDITIONS: Mild Cognitive Impairment; Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Low dose (Experimental)
  Interventions: Drug: grape seed polyphenolic extract, resveratrol
- moderate dose (Experimental)
  Interventions: Drug: grape seed polyphenolic extract, resveratrol
- High dose (Experimental)
  Interventions: Drug: grape seed polyphenolic extract, resveratrol

INTERVENTIONS:
Drug: grape seed polyphenolic extract, resveratrol — Bioactive Dietary Polyphenol Preparation (BDPP) is a combination of two nutraceutical preparations (grape seed polyphenolic extract [GSE], and resveratrol) that contain abundant concentrations of polyphenols.
  Other Names: Bioactive Dietary Polyphenol Preparation

SUMMARY:
Mild Cognitive Impairment (MCI) represents a group of persons who are at risk of incident dementia in the near-term. Persons with MCI who have deficits in short-term recall (amnestic MCI) are at significant risk of incident Alzheimer's disease (AD) (termed prodromal AD), and thus represent a worthy target for secondary prevention interventions.

There is increasing evidence that risk factors for metabolic syndrome (such as prediabetes and type 2 diabetes) increase risk of incident cognitive impairment and possibly AD, and evidence that the neurons of the AD brain are in fact insulin resistant with diminished glucose uptake under physiological conditions. Thus, persons with MCI and prediabetes or type 2 diabetes may be at particular risk of incident cognitive impairment and AD.

A large clinical trial (ACCORD)1 demonstrated that tight control of peripheral blood glucose does not improve cognitive (or other health) outcomes in older persons with peripheral insulin resistance. Thus, there is a need to target cognitive outcomes in persons with MCI and metabolic risk factors, and a drug targeting insulin resistance with good blood-brain-barrier (BBB) penetrance can potentially accomplish these objectives. While there is a phase III study of intranasal insulin targeting this strategy, nutraceuticals offer a low-tech solution that would be more suitable to future secondary prevention trials in MCI.

Bioactive Dietary Polyphenol Preparation (BDPP) is a combination of two nutraceutical preparations grape seed polyphenolic extract (GSE), and resveratrol that contain abundant concentrations of polyphenols. The investigators have found that oral BDPP administration was associated with improved cognition and brain plasticity long-term potentiation (LTP) in mouse models of metabolic syndrome and AD, as well as lowering brain amyloid and tau burden in an AD mouse model2-4. The investigators have demonstrated excellent absorption of oral BDPP in a small study in humans and similarly excellent CSF penetration of oral BDPP in rats, but it is crucial to demonstrate safety and CSF penetration of oral BDPP in humans to assess its potential as a treatment for MCI and prediabetes or type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-90 years inclusive
* Amnestic MCI
* Impaired fasting glucose (IFG), defined by American Diabetes Association criteria (fasting blood sugar between 100 and 125 mg/dl) or clinically stable type 2 diabetes
* Knowledgeable informant (KI) who spends at least 5 hours/week with the participant and can provide information about the participant's psychosocial functioning

Exclusion Criteria:

* Deemed too unstable medically or neurologically to safely enroll in trial of research medication
* Type 1 Diabetes Mellitus
* Diagnosis of dementia due to Alzheimer's disease

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-06; Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Assessment of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 4 months
Confirm brain penetrance of BDPP by measuring levels of BDPP constituents in cerebrospinal fluid (CSF). | 4 months
Evaluate BDPP effect on mood with Neuropsychiatric Inventory and Cornell Scale for Depression in Dementia. | 4 months
Evaluate BDPP effect on cognition with measures of memory, executive function, and attention measures (composite) | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Roserberg, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States